CLINICAL TRIAL: NCT02689193
Title: IDIS Project Work Package 2: Establishing a Biobank at ITM and Collaborating Centres
Acronym: IDIS
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Sihanouk Hospital Center of HOPE (Other); Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other); Vlaams Instituut voor Biotechnologie (Unknown)
Responsible Party: Sponsor
Other Study IDs: IDIS
Record Dates: First submitted 2016-01-29; First posted 2016-02-23 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Salmonella Septicemia; Salmonella Infections; Fever; Blood Stream Infections; Parasitic Infections
Keywords: Proteomics; Rapid Diagnostic Test; Salmonellosis
MeSH Terms: conditions — Salmonella Infections; Fever; Parasitic Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, plasma, serum and urine.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Salmonella: Patients for whom blood cultures grew Salmonella species.
  Interventions: Other: Blood sampling
- No pathogen: Patients for whom blood cultures did not grow a pathogen and no pathogen was detected using other routine care diagnostics (e.g. malaria with the use of a malaria rapid test).
  Interventions: Other: Blood sampling
- Another pathogen: Patients for whom blood cultures grew with another pathogen or a pathogen was detected using other routine care diagnostics (e.g. malaria with the use of malaria rapid test).
  Interventions: Other: Blood sampling
- Healthy controls: Healthy controls. Patients without fever but from whom blood is drawn for another reason (e.g. check of cholesterol).
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Blood sampling (Volume depending on age, minimum 2.0 ml, maximum 10.9 ml extra)

SUMMARY:
The IDIS study aims to develop a new rapid diagnostic test for invasive salmonellosis using samples (blood, urine) collected from patients with fever and healthy controls at the Institute of Tropical Medicine (ITM) and collaborating centers. The samples are collected after informed consent and/or assent is given by the participant and are stored in a -80 ⁰C freezer after processing (centrifugation and/or aliquoting). Basic information regarding the patient and the samples are coded and stored in a protected Microsoft Access database. The samples will be shipped to Belgium for proteomic analysis. Identification of Salmonella specific proteins in the samples will hopefully support the development of a rapid diagnostic test. Once this test has been developed, the samples will also be used for validation and evaluation of this test.

DETAILED DESCRIPTION:
The aim of the project is the identification of Salmonella specific proteins that can be detected in samples derived from the host (= humans) during an acute infection. This can support the development of rapid tests to improve the diagnosis of invasive Salmonellosis.

The study is taking place at the travel clinic of the Institute of Tropical Medicine in Antwerp, Belgium, and at the Sihanouk Hospital Center of HOPE in Phnom Penh, Cambodia. It is planned to start in 2016 at the Centre Hospitalier de Kingasani in Kinshasa, Democratic Republic of the Congo in collaboration with the Institut National de Recherche Biomédicale in Kinshasa, Democratic Republic of the Congo. The expected number of participants in total is 2500.

Patients (children and/or adults) presenting with (a history of) fever are asked permission (informed consent and/or assent) to draw additional blood samples (along with routine care samples, so no need for additional venipuncture), and for the long term storage of these samples (whole blood and plasma) in a freezer together with left-over serum and urine samples. They are also asked permission for the collection of coded data including basic demographic, clinical and laboratory data.

Blood for plasma and urine are centrifugated. All samples are aliquoted into cryotubes (coded labelling) before storage in a -80 ⁰C freezer.

Depending on the final diagnosis, patients can be divided in 4 groups:

1. Patients for whom blood cultures grew Salmonella species
2. Patients for whom blood cultures did not grow a pathogen
3. Patients for whom blood cultures grew with another pathogen
4. Healthy controls

The frozen samples collected in Cambodia and the Democratic Republic of the Congo will be shipped to Belgium.

All selection of all the samples collected will undergo proteomic analysis by researchers of the Institute of Tropical Medicine in collaboration with the Vlaams Instituut voor Biotechnologie and coded data related to the samples is shared with these partners.

Once this test has been developed, the samples will also be used for validation and evaluation of this test.

ELIGIBILITY:
A. Travel clinic Institute of Tropical Medicine (ITM) Antwerp

Inclusion Criteria:

Adults (≥ 18 years) and children aged 3 years to 18 years with (suspicion of) fever and:

1. presenting at ITM travel clinic with history of fever (axillary T° ≥ 38°C) and/or chills/rigor and sweats within 3 days prior to consultation
2. presenting at ITM travel clinic for routine check-up ("apparently healthy")
3. with recent (< 2 weeks) stay in tropical country

Exclusion Criteria:

Refusal to participate

B. Sihanouk Hospital Center of HOPE (SHCH)

Inclusion Criteria:

Adults (≥ 18 years) with (suspicion of) fever and:

1. Presenting at the in- and outpatient department of SHCH with a history of fever (axillary T≥ 38°C) and/or/chills/rigor and sweats within 3 days prior to consultation

Exclusion Criteria:

1. Refusal to participate
2. Not able to give informed consent

Inclusion Criteria:

Adults (≥ 18 years) and children aged 2 months to 18 years with (suspicion of) fever and:

1. Blood culture request by treating physician

Exclusion Criteria:

1. Not able or willing to give informed consent
2. A hemoglobin level that is considered too low for weight and age

Inclusion Criteria:

Adults (≥ 18 years) and children aged 2 months to 18 years with (suspicion of) fever and:

1. Blood culture request by treating physician

Exclusion Criteria:

1. Not able or willing to give informed consent
2. A hemoglobin level that is considered too low for weight and age

Min Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults presenting with (a history of) fever and healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2014-09; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Detection of bacterial proteins through Selected Reaction Monitoring (SRM) measured in the unit m/z | 2 years
  Detection of bacterial proteins in the collected urine and blood samples through Selected Reaction Monitoring (SRM) measured in the unit m/z (whereby m = the atomic mass and z = the charge of the ion)
Quantification of bacterial proteins measured through Selected Reaction Monitoring (SRM) as ion counts | 2 years
  Quantification of bacterial proteins measured through Selected Reaction Monitoring (SRM) as ion counts in the collected urine and blood samples
Ranking of detected bacterial proteins based on detection per number of samples and on ion counts | 2 years
  Ranking of detected bacterial proteins based on:
  * Detection of bacterial proteins per number of Salmonella positive and Salmonella negative urine and blood samples
  * Protein abundance measured as ion counts
Colorimetric detection of the selected proteins by ELISA measured in the unit optical density | 2 years
  Colorimetric detection of the selected proteins by ELISA measured in the unit optical density (OD) and expressed as percentage present in Salmonella positive and Salmonella negative urine and blood samples
Integration of the selected proteins into a rapid diagnostic test based on a lateral flow format | 4 years
Evaluation of the test expressed as percentage positive in samples | 4 years
  Evaluation of the test on the collected blood and urine samples expressed as percentage positive in Salmonella positive and Salmonella negative samples

CONTACTS AND LOCATIONS:
Overall Officials: Laura Kuijpers, MD, MSc, Principal Investigator — Institute of Tropical Medicine, Antwerp, Belgium; Panha Chung, Principal Investigator — Sihanouk Hospital Center of HOPE (SHCH), Phnom Penh, Cambodia; Ange Landela, MD, Principal Investigator — Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo
Locations (3):
- Institute of Tropical Medicine, Antwerp, Flanders, Belgium
- Sihanouk Hospital Center of Hope (SHCH), Phnom Penh, Cambodia
- Institut National de Recherche Biomédicale, Kinshasa, Democratic Republic of the Congo